CLINICAL TRIAL: NCT01590407
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 3-Part Study of Orally Administered ALS-002200 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Dosing and Food-effect in Healthy Volunteers, and Multiple Ascending Dosing in Subjects With Chronic Hepatitis C Genotype 1 Infection
Brief Title: First in Human Study of ALS-002200; Single Dose, Food Effect in Healthy Volunteers; Multiple Doses in Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALS-2200-101
Record Dates: First submitted 2012-03-12; First posted 2012-05-03 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- ALS-002200 (Experimental)
  Interventions: Drug: ALS-002200
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALS-002200 — ALS-002200
  Arms: ALS-002200
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, 3-part study will assess the safety, tolerability, and pharmacokinetics of orally administered ALS-002200 in healthy volunteers (HV) and subjects with chronic hepatitis C (CHC) genotype 1 infection.

Part 1 will assess single ascending dosing pharmacokinetics and safety in HV. Part 2 will assess food effects on pharmacokinetics in HV. Part 3 will assess multiple ascending dosing pharmacokinetics and safety in subjects with CHC genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent.
* In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned.
* Subject is in good health as deemed by the investigator.
* Creatinine clearance of greater than 50 mL/min (Cockcroft-Gault)
* Male or female, 18-55 years of age for HV and 18-65 years of age for subjects with CHC.
* Body mass index (BMI) 18-32 kg/m2 inclusive for HV and 18-36 kg/m2 for subjects with CHC, minimum weight 50 kg in both populations.
* A female is eligible to participate in this study if she is of non childbearing potential.
* If male, subject is surgically sterile or practicing specific forms of birth control.

Additional inclusion criteria for subjects with CHC genotype 1 infection:

* Positive HCV antibody and a positive HCV RNA at screening.
* Documentation of CHC infection for greater than 6 months at screening
* CHC genotype 1 infection at screening
* HCV RNA viral load ≥ 105 and ≤108 IU/mL using a sensitive quantitative assay.
* Liver biopsy within two years or Fibroscan evaluation within 6 months prior to screening that clearly excludes cirrhosis. Fibroscan liver stiffness score must be < 12 kPa.
* Absence of hepatocellular carcinoma as indicated by an ultrasound scan conducted during screening
* No prior treatment for CHC
* Absence of history of clinical hepatic decompensation.
* Laboratory values include:

  * Prothrombin time < 1.5x ULN
  * Platelets > 120,000/mm3
  * Albumin > 3.5 g/dL, bilirubin < 1.5 mg/dL at screening (subjects with documented Gilbert's disease allowed).
  * Serum alanine aminotransferase (ALT) concentration < 5 x ULN
  * Alpha Fetoprotein (AFP) concentrations ≤ ULN. If AFP is ≥ ULN, absence of a hepatic mass must be demonstrated by ultrasound within the screening period.

Exclusion Criteria:

* Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder.
* Positive test for HAV IgM, HBsAg, HCV Ab (HV only), or HIV Ab.
* Abnormal screening laboratory results that are considered clinically significant by the investigator.
* Drug allergy such as, but not limited to, sulfonamides and penicillins, including those experienced in previous trials with experimental drugs.
* Participation in an investigational drug trial or having received an investigational vaccine within 30 days or 5 half lives (whichever is longer) prior to study medication.
* Clinically significant blood loss or elective blood donation of significant volume.
* For healthy subjects, history of regular use of tobacco.
* The subject has a positive pre-study drug screen.
* Laboratory abnormalities including:

  * Thyroid Stimulating Hormone (TSH) > ULN
  * Hematocrit < 34 %
  * White blood cell counts < 3,500/mm3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-12-31 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2013-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to Day 31
  data points measured include patient reported adverse events, physical exams, vital signs, 12-lead ECGs and clinical lab results

SECONDARY OUTCOMES:
Cmax | pre-dose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 240 hours post dose
AUC | pre-dose and 0.25, 0.5, 1, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 240 hours post dose
HCV ribonucleic acid (RNA) viral load reduction | Baseline to Day 31
Amino Acid Changes in HCV polymerase NS5b | Baseline up to Month 6
  Comparison of baseline with on-treatment or post-treatment Hepatitis C virus (HCV) NS5B RNA sequence

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Biotrial, Rennes, Brittany Region
  - Biotrial, Paris
- Arensia, Chisinau, Moldova
- Arensia, Bucharest, Romania